CLINICAL TRIAL: NCT02110030
Title: Effectiveness of Two Electrotherapy Techniques to Treat Subacromial Impingement Syndrome
Acronym: TENSIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Collaborators: Public Health Service of Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCJC-13
Record Dates: First submitted 2014-04-04; First posted 2014-04-10 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Transcutaneous electrical nerve stimulation (TENS); Ultrasound; Interferential current therapy; Rehabilitation; Shoulder pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcutaneous nerve stimulation (Experimental): The group with transcutaneous nerve stimulation (TENS) received electrical stimulation for 15 sessions at a frequency of 80 Hz and with a pulse width of 150 ns.
  The group with TENS received electrical stimulation by using an approved electrotherapy device (Endomed 182, Enraf-nonius, Germany). The TENS was applied by using 4 surface electrodes (5x5 cm Prim-Trode, Spain) into two channels: supraspinatus fossa and the insertion of the rotator cuff (channel 1) and "V" deltoid " (channel 2).
  Interventions: Device: Transcutaneous nerve stimulation
- Interferential Currents (Active Comparator): The group with Interferential Currents (IC) received a base frequency of 4000 Hz by using the same approved electrotherapy device than the TENS group (Endomed 182, Enraf-nonius, Germany).
  Interventions: Device: Interferential Currents

INTERVENTIONS:
Device: Transcutaneous nerve stimulation — The group with TENS received electrical stimulation (Endomed 182, Enraf-nonius, Germany) at a frequency of 80 Hz and with a pulse width of 150 ns. The TENS was applied by using 4 surface electrodes (5x5 cm Prim-Trode, Spain) into two channels: supraspinatus fossa and the insertion of the rotator cuff (channel 1) and "V" deltoid " (channel 2). The current intensity was set 3 times during each session according to each patient's sensitivity. Current was strong but it did not exceed the threshold of pain.
  Other Names: TENS
  Arms: Transcutaneous nerve stimulation
Device: Interferential Currents — The group with IC received a base frequency of 4000 Hz (Endomed 182, Enraf-nonius, Germany) with an amplitude-modulated frequency (AMF) and slope of 1/1 in tetrapolar mode, as previously indicated. For IC, the same number and type of surface electrodes (5x5 cm Prim-Trode, Spain) were placed onto the anterior and posterior deltoid, supraspinatus fossa and "V" deltoid. Similarly, the intensity of the current was set 3 times per session and the stimulation was strong but comfortable (without exceeding the threshold of pain).
  Other Names: IC
  Arms: Interferential Currents

SUMMARY:
Objective: The investigators aimed to compare the effectiveness of transcutaneous electrical nerve stimulation (TENS) and interferential currents (IC) to improve shoulder functionality and to reduce perceived pain in patients with subacromial impingement syndrome (SIS). Design: Thirty-six patients with unilateral shoulder pain and diagnosed as having SIS were randomly assigned into two groups: TENS (n=18; 51±7 years) and IC (n=18; 47±6 years). Patients in both groups received fifteen 30-min sessions of the assigned treatment for a period of 3 weeks. Before and after the treatment, shoulder pain was measured using a 100-mm visual analog scale and shoulder functionality was measured using the Constant-Murley scale.

DETAILED DESCRIPTION:
Subjects

The subjects for this study were recruited from a waiting list from patients with acute shoulder pain at the Almendrales Medicine and Physiotherapy Center (Madrid, Spain). To be included in the list they had to be older than 18 years and have had unilateral shoulder pain for more than 1 month. Potential participants were then examined by an independent specialist and the diagnosis of SIS was made according to the Hawkins and Jobe tests. The use of X-ray, ultrasonography and magnetic resonance imaging permitted objective diagnoses of SIS and the exclusion of patients with other shoulder pathologies. With these inclusion criteria, a total of 63 patients were recruited for the experiment. The following participants were excluded from the investigation: individuals with rotator cuff tears or calcification; individuals with the presence of acute trauma; patients who were receiving treatment for their SIS with another method; patients with previous surgery or intra-articular injections; individuals with contraindications against electrotherapy. Ethical approval for this experiment was previously obtained by the local Institutional Review and all participants signed an informed consent prior to enrolling in the investigation.

Treatment groups

The experimental design was a randomized and double-blind clinical trial. After preliminary examination, the patients were randomly assigned into two groups: transcutaneous electrical nerve stimulation (TENS) and interferential currents (IC). A set of sealed and sequentially numbered opaque envelopes was used for group assignment. The study was double-blind because the examiner had no contact with the patient during the duration of the treatment and patients were not informed about the electrotherapy technique they received during the investigation.

Intervention

For both experimental groups, the treatments were applied over a period of 3 weeks, including a total of 15 sessions (approximately 5 sessions per week). In each session, the electrical stimulation technique was administered for 30 minutes while the subjects were comfortable seated in an adjustable chair. The group with TENS received electrical stimulation (Endomed 182, Enraf-nonius, Germany) at a frequency of 80 Hz and with a pulse width of 150 ns. The TENS was applied by using 4 surface electrodes (5x5 cm Prim-Trode, Spain) into two channels: supraspinatus fossa and the insertion of the rotator cuff (channel 1) and "V" deltoid " (channel 2). The current intensity was set 3 times during each session according to each patient's sensitivity. Current was strong but it did not exceed the threshold of pain. The group with IC received a base frequency of 4000 Hz (Endomed 182, Enraf-nonius, Germany) with an amplitude-modulated frequency (AMF) and slope of 1/1 in tetrapolar mode, as previously indicated. For IC, the same number and type of surface electrodes (5x5 cm Prim-Trode, Spain) were placed onto the anterior and posterior deltoid, supraspinatus fossa and "V" deltoid. Similarly, the intensity of the current was set 3 times per session and the stimulation was strong but comfortable (without exceeding the threshold of pain). The treatments were administered by an experienced physiotherapist blinded to the aim of this investigation.

Outcome measurements

Shoulder pain was evaluated before and the day after the end of treatments by using a 100 mm visual analog pain scale. Functional status in the shoulder joint was evaluated two days before, after 8 sessions of treatment and the day after the end of the treatment by using the Constant-Murley scale. This scale is valid to assess the overall functionality of a normal, a diseased or a treated shoulder. In this scale, 35% of the total value was allocated from subjective assessments of pain (20%) and self-evaluation of activities of daily living (15%; including shoulder pain during sleeping, dysfunction during free time or sports and dysfunction during working activities). The remaining 65% of the total value came from objective measures of range of movement and shoulder strength. Within the objective evaluation, the range of motion during internal and external rotation, arm flexion and lateral elevation (all measured by using an inclinometer) amounted to 10% each of the total score. Strength was measured using the muscular balance system by Daniels30 and counted for 25% of the total score. Thus, a young and healthy patient can have a maximal punctuation of 100 points. The pre-to-post treatment shoulder evaluation was performed by the same independent experimenter using the same instruments. This experimenter was blinded to the treatment assigned to each participant.

Statistical analysis

All the data were analyzed using SPSS v.20 statistical package. Descriptive statistics were calculated for each group (mean and standard deviation). Normality was tested with the Shapiro-Wilk test. All the variables presented a normal distribution in this test (P > 0.05). Baseline characteristics were compared using the analysis of variance (ANOVA) for measuring independent data. Pre-to-post treatment data and the comparison between groups were performed by using two-way ANOVA (group x time). After a significant F test, differences between means were identified using Tukey's HSD post hoc procedure. The level of significance was established at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* The subjects for this study were recruited from a waiting list from patients with acute shoulder pain at the Almendrales Medicine and Physiotherapy Center (Madrid, Spain).
* To be included in the list they had to be older than 18 years and have had unilateral shoulder pain for more than 1 month.
* Potential participants were then examined by an independent specialist and the diagnosis of SIS was made according to the Hawkins and Jobe tests.
* The use of X-ray, ultrasonography and magnetic resonance imaging permitted objective diagnoses of shoulder impingement syndrome and the exclusion of patients with other shoulder pathologies.

Exclusion Criteria:

* The following participants were excluded from the investigation: individuals with rotator cuff tears or calcification; individuals with the presence of acute trauma; patients who were receiving treatment for their shoulder pain with another method; patients with previous surgery or intra-articular injections; individuals with contraindications against electrotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Shoulder functionality | Before and after the 3 weeks of electrotherpy treatment
  Functional status in the shoulder joint was evaluated by using the Constant-Murley scale. This scale is valid to assess the overall functionality of a normal, a diseased or a treated shoulder. In this scale, 35% of the total value was allocated from subjective assessments of pain (20%) and self-evaluation of activities of daily living (15%; including shoulder pain during sleeping, dysfunction during free time or sports and dysfunction during working activities). The remaining 65% of the total value came from objective measures of range of movement and shoulder strength.
  Shoulder functionality was measured by using a 0-100 point scale.
  The pre-to-post treatment shoulder evaluation was performed by the same independent experimenter using the same instruments.
Shoulder pain | Before and after the 3 weeks of electrotherpy treatment
  Shoulder pain was evaluated before and the day after the end of treatments by using a 100 mm visual analog pain scale.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Del Coso, PhD, Principal Investigator — Camilo Jose Cela University
Locations (1):
- Health Center Almendrales, Madrid, Spain

REFERENCES:
- [Background] Constant CR, Gerber C, Emery RJ, Sojbjerg JO, Gohlke F, Boileau P. A review of the Constant score: modifications and guidelines for its use. J Shoulder Elbow Surg. 2008 Mar-Apr;17(2):355-61. doi: 10.1016/j.jse.2007.06.022. Epub 2008 Jan 22. No abstract available. PMID 18218327